CLINICAL TRIAL: NCT03462823
Title: Randomized Controlled Trial for the Use of an Osteoconductive Scaffold in ACL-Reconstruction
Brief Title: Use of an Osteoconductive Scaffold in ACL-Reconstruction
Acronym: ACLROCS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sandro Fucentese (Other)
Responsible Party: Sponsor-Investigator, Sandro Fucentese, Head of Knee Surgery, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W652
Record Dates: First submitted 2017-12-29; First posted 2018-03-13 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture; ACL; ACL Injury
Keywords: ACL Reconstruction; Osteoconductive Scaffold; Bone Tunnel Widening
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Randomized patient-blinded two-group parallel comparison trial using an active comparator.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control treatment (Active Comparator): ACL-reconstruction using hamstring autograft with hybrid fixation in accordance with in-house standard of care.
  Interventions: Device: Hamstring tendon-only repair
- Experimental treatment (Experimental): ACL-reconstruction using hamstring autograft with hybrid fixation combined with the osteoconductive device under study.
  Interventions: Device: Osteoconductive scaffold-hamstring tendon composite repair

INTERVENTIONS:
Device: Osteoconductive scaffold-hamstring tendon composite repair — The device under study is a composite bone substitute composed of a natural mineral matrix of bovine origin, reinforced with biodegradable synthetic polymers and natural collagen derivatives of bovine origin (smartbone, IBI S.A., Switzerland).
  Arms: Experimental treatment
Device: Hamstring tendon-only repair — ACL-reconstruction using hamstring autograft with hybrid fixation in accordance with in-house standard of care.
  Arms: Control treatment

SUMMARY:
Primary objective of the study is to evaluate efficacy of the surgical technique for ACL reconstruction using an osteoconductive scaffold, enlaced into the hamstring tendon autograft, compared to the traditional technique.

DETAILED DESCRIPTION:
Reconstruction of the anterior cruciate ligament (ACL) using autograft tissue is currently recommended as the standard of care following an ACL tear or rupture, with the bone-tendon-bone (BTB) graft and hamstring tendon graft the most common. Although a BTB autograft is widely recognized to offer high mechanical performance and rapid graft healing, these advantages come at the cost of a longer surgery time and higher risk of severe patient discomfort at the graft harvest site. Use of a hamstring tendon autograft is less painful, but is generally slower to heal with higher risk of mechanical graft failure due to poor bone ingrowth. The aim of the current study is to augment graft-to-bone incorporation by use of an osteoconductive scaffold enlaced into the hamstring tendon autograft. This bovine derived composite bone substitute is inserted into the articular aperture of the femoral bone tunnel and should provide an osteoconductive / osteoinductive environment at a biomimetic attachment site leading to improved secondary graft-fixation and a reduced incidence of tunnel widening.

Primary objective of the study is to evaluate efficacy of the surgical technique for ACL reconstruction using an osteoconductive scaffold, enlaced into the hamstring tendon autograft, compared to the traditional technique.

Secondary objectives aim to assess the clinical outcome of the interventional treatment including patient subjective knee function and objective measures of knee stability.

ELIGIBILITY:
Inclusion

* Acute unilateral complete tear of the ACL that occurred within 18 weeks before planned surgery and requires reconstruction of the
* Informed consent as documented by signature

Exclusion Criteria:

* Prior ACL reconstruction or other surgical procedure on the affected knee.
* Prior fracture of the affected leg.
* Multi-ligament reconstruction.
* Previous or current ACL injury on contra-lateral leg.
* Medical condition or comorbidity that would interfere with study participation.
* The patient is mentally compromised.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Other clinically significant concomitant disease states (e.g. renal failure, hepatic dysfunction, cardiovascular disease, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-04-29 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Bone tunnel volume | 0, 4.5, 12 months post surgery
  CT based relative change of the femoral bone tunnel volume from baseline to follow-up 1 and 2.

SECONDARY OUTCOMES:
IKDC Subjective Knee Evaluation Form | 0 and 42 days, 6 months, 1, 2 and 5 years post surgery
  International Knee Documentation Committee Subjective Knee Evaluation Form is designed to detect improvement or deterioration in symptoms, function and sports activities due to knee impairment for patients with a variety of knee conditions including ligament injuries. It is a patient-completed questionnaire available in multiple languages including German with an ordinal scoring system ranging from 0 (highest level of symptoms or lowest level of function) to 100 (no limitation with daily or sporting activities and the absence of symptoms).
Lysholm Knee Scoring Scale | 0 and 42 days, 6 months, 1, 2 and 5 years post surgery
  To evaluate outcomes of knee ligament surgery, particularly symptoms of instability. It has an ordinal scoring system ranging from 0 to 100 (No symptoms or disability). A validated German version will be used.
Tegner Activity Scale | 0 and 42 days, 6 months, 1, 2 and 5 years post surgery
  The Tegner activity scale (TAS) is used to measure the change in physical activity from pre-injury to follow-up. Patient's activity is scored on a scale with 11 levels from level 0 (on sick leave/disability) to level 10 (participation in competitive sports such as soccer at a national or international elite level). Evaluated will be the difference in score from pre-injury (assessed at baseline visit) to follow-up.
KT-1000 Arthrometer Test | 0 and 42 days, 6 months, 1, 2 and 5 years post surgery
  The KT-1000 Arthrometer Test measures anterior displacement of the tibial plateau on the femur at a specific force. Its output variable is defined as the difference in full millimeters between the tibial displacement of the ACL reconstructed knee and the normal contralateral side.
Lachmann Test | 0 and 42 days, 6 months, 1, 2 and 5 years post surgery
  The Lachman test measures anterior displacement conducted manually by the clinician. It is graded as the difference from the normal contralateral side as 0 (<3 mm), 1 (3 to 5 mm), or 2 (>5 mm).
Pivot shift test | 0 and 42 days, 6 months, 1, 2 and 5 years post surgery
  The pivot shift test assesses the combined tibio-femoral rotation and anterior tibial translation. The pathologic motion elicited is graded as a glide (grade 1), clunk (grade 2), or gross clunk with locking (grade 3). A normal finding is graded as zero. The outcome measure is calculated from the difference between affected (repaired) and intact knee.
Bone tunnel width | 0 and 42 days, 12 and 24 months post surgery
  Bone tunnel width will additionally be assessed on plain radiograph. Standard posteroanterior radiographs of the knee in full extension will be used. Bone tunnel width will be assessed at the widest part of the femoral bone tunnel. Assessed will be the relative change in femoral bone tunnel width.
Osteoconductive scaffold-bone integration | day 0, 4.5 and 12 months post surgery
  For a quantitative analysis of Osteoconductive scaffold (OCS)-bone integration, the mineral density profile along a predefined line will be examined. A slice showing the central portion of the OCS in the axial plane will be selected. A straight line of 2 cm length will be drawn perpendicular to the long axis of the OCS using image analysis software (Mimics). The CT-values along this line will be recorded and evaluated in the following way. Since the CT-values change according to the bone mineral density, the profile along the line will have a minimum at the interface of the tunnel wall and the OCS and a maximum on the OCS. The difference in Hounsfield units from the cancellous bone in the tunnel wall and the OCS-bone interface will be used as a measure for the degree of osseous integration of the implant.

OTHER OUTCOMES:
Patient safety | 0 and 42 days, 6 months, 1, 2 and 5 years post surgery
  Any occurrence of intra-operative complications will be recorded on the case report forms. Post-operative (serious) adverse events will be recorded at each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Fucentese, Principal Investigator — Head of Knee Surgery
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gotschi T, Hodel S, Kuhne N, Bachmann E, Li X, Zimmermann SM, Snedeker JG, Fucentese SF. Osteoconductive Scaffold Placed at the Femoral Tunnel Aperture in Hamstring Tendon ACL Reconstruction: A Randomized Controlled Trial. Orthop J Sports Med. 2023 Jun 5;11(6):23259671231174478. doi: 10.1177/23259671231174478. eCollection 2023 Jun. PMID 37347015

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT03462823/Prot_SAP_000.pdf